CLINICAL TRIAL: NCT07391228
Title: Cognitive Alterations in Pulmonary Arterial Hypertension (PAH): an Exploratory Cross- Sectional Study
Brief Title: Cognitive Alterations in Pulmonary Arterial Hypertension (PAH)
Acronym: COG-PAH
Status: Active, not recruiting | Type: Observational
Sponsor: Alessandra Gorini (Other)
Responsible Party: Sponsor-Investigator, Alessandra Gorini, Professor Alessandra Gorini, PhD, Psychologist, Neuropsichology, Psychotherapist, Istituti Clinici Scientifici Maugeri SpA
Organization: Istituti Clinici Scientifici Maugeri SpA (Other)
Other Study IDs: COG-PAH - CTSM180-25
Record Dates: First submitted 2025-11-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Cognitive Functions; Neuropsychological Assessment; Cross-sectional Study
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAH patients: The first group is composed by patients over 18 years with a confirmed diagnosis of PAH, which are clinically stable (according to the treating physician's judgement) and have no neurological and psychiatric comorbidities
- Healthy subjects: Healthy controls matched for age (± 3 years), gender, handedness and educational level, with no current or past organic and/or psychiatric disorders

SUMMARY:
Pulmonary Arterial Hypertension (PAH) is a rare chronic disease marked by a pathological and sustained increase in pulmonary artery pressure as a result of structural and functional changes within the pulmonary vasculature. Beyond its cardiopulmonary manifestations, a growing body of evidence suggests that PAH may also affect cerebral hemodynamics and cognitive functioning as a consequence of prolonged reductions in cerebrovascular oxygenation potentially underlying the frontal-executive, attentional, and mnestic impairments reported in this population. Despite these preliminary findings, the few studies currently available have significant methodological limitations, such as the lack of appropriate control groups or the inclusion of other pulmonary hypertension subtypes in the cohort. In addition, they tend to rely on global cognitive screening tests that are unsuitable for the precise characterization of domain-specific alterations, such as those observed in PAH.

This study aims to address these limitations by employing a battery of computerized neuropsychological tests to detect the presence of selective cognitive alterations in individuals diagnosed with PAH, through comparison with a control group matched for age, sex, handedness and schooling.

The project is designed as a cross-sectional observational study conducted at a single center, with the primary aim to assess the presence of selective cognitive alterations in patients diagnosed with PAH, comparing their performance with that of a healthy control group matched for age, sex, handedness, and level of education.

The secondary objective is to explore the relationship between cognitive variables and clinical variables in patients with PAH, such as disease duration, age at diagnosis, oxygen therapy, and reported comorbidities.

Participants will be assessed in a single in-person session at the IRCCS Maugeri Milano, using a computerised battery of tests that will last approximately 50 minutes.

Recruitment will take place consecutively among patients hospitalised at the U.O. Rehabilitative Cardiology of the IRCCS Maugeri- Milano Via Camaldoli. Healthy controls will be identified on a voluntary basis among IRCCS Maugeri staff, healthy family members of patients, or through other authorised internal channels.The total duration of the study is expected to be 24 months, with an estimated start date of 15/11/2025 and end date of 31/07/2027.

Participants will undergo an initial collection of medical history data to verify their eligibility for the study. The information collected will include sociodemographic data (sex, age, marital status, number of children, employment status, level of education, years of schooling) and clinical data (past and recent medical history, current drug therapies, behavioural habits such as smoking and/or alcohol consumption, handedness). Data relating to performance in neuropsychological tests will be collected using the Inquisit 7.0 by Millisecond platform (https://www.millisecond.com/). Cognitive tasks will be performed individually and in person on an HP Envy x360 PC running Windows 11.

Assessment tools Neuropsychological tests were chosen to investigate selective alterations in cognitive functions related to brain areas whose activation was found to be altered in PAH patients in the aforementioned studies, such as the selective and sustained attention, working memory, processing speed and cognitive flexibility, inhibitory control, interference contrast, categorical abstraction, as well as learning and long-term verbal memory.

Selected test are listed below:

* Iowa Gambling Task (IGT): developed by Bechara and colleagues (1994);
* Emotional Stroop Task (EST): a variant of the classic Stroop Test, developed by Smith and Waterman (2003);
* The Rey Auditory Verbal Learning Test (RAVLT): validated in the Italian version by Carlesimo et al., (1995); The Visual Simon Task (VST): a variant of the Simon Task (2004); The Wisconsin Card Sorting Test (WCST): by Heaton et al., (1993);

DETAILED DESCRIPTION:
Background Pulmonary Arterial Hypertension (PAH) is a rare chronic disease marked by a pathological and sustained increase in pulmonary artery pressure as a result of structural and functional changes within the pulmonary vasculature, such as vasoconstriction, vascular remodeling, inflammation, and endothelial dysfunction. Over time, these processes lead to a progressive increase in pulmonary vascular resistance and consequent right ventricular overload, which gradually results in hypertrophy, dilatation, right ventricular failure, and ultimately heart failure.

Beyond its cardiopulmonary manifestations, a growing body of evidence suggests that PAH may also affect cerebral hemodynamics and cognitive functioning as a consequence of prolonged reductions in cerebrovascular oxygenation. Findings from brain imaging studies indicate structural changes in patients with PAH, characterized by reduced gray matter volume in regions associated with cognitive, autonomic, and emotional regulation, such as the hippocampus, amygdala, cerebellum, insula, thalamus, and temporal, frontal, occipital, and cingulate cortices.

These alterations likely reflect chronic brain tissue damage caused by prolonged hypoxic- ischemic conditions, potentially underlying the frontal-executive, attentional, and mnestic impairments reported in this population.

Despite these preliminary findings, the few studies currently available have significant methodological limitations, such as the lack of appropriate control groups or the inclusion of other pulmonary hypertension subtypes in the cohort. In addition, they rely on global cognitive screening tests, which are unsuitable for the precise characterization of domain-specific alterations, such as those observed in PAH.

This study aims to address these limitations by employing a battery of computerized neuropsychological tests to detect the presence of selective cognitive alterations in individuals diagnosed with PAH, through comparison with a control group matched for age, sex, handedness and schooling.

* Primary objective To assess the presence of selective cognitive alterations in patients diagnosed with PAH, comparing their performance with that of a healthy control group matched for age, sex, handedness and level of education.
* Secondary objective To explore the relationship between cognitive variables and clinical variables in patients with PAH, such as disease duration, age at diagnosis, oxygen therapy, and reported comorbidities.

Design of the study The project is designed as a cross-sectional observational study conducted at a single centre. No intervention other than normal clinical practice is planned.

Participants will be assessed in a single in-person session at the IRCCS Maugeri Milano, using a computerised battery of tests that will last approximately 50 minutes.

Recruitment will take place consecutively among patients hospitalised at the U.O. Rehabilitative Cardiology of the IRCCS Maugeri- Milano Via Camaldoli. Healthy controls will be identified on a voluntary basis among IRCCS Maugeri staff, healthy family members of patients, or through other authorised internal channels.

The total duration of the study is expected to be 24 months, with an estimated start date of 15/11/2025 and end date of 31/07/2027. The start date may be subject to change depending on the approval times of the relevant Ethics Committee.

The protocol includes the following operational phases:

* Definition, preparation and programming of scripts for the administration of neuropsychological tests;
* Selection and enrollment of the sample and administration of the test battery;
* Data analysis and dissemination of results.

Material and methods Data collection platform Participants will undergo an initial collection of medical history data to verify their eligibility for the study. The information collected will include sociodemographic data (sex, age, marital status, number of children, employment status, years of schooling) and clinical data (past and recent medical history, current drug therapies, behavioural habits such as smoking and/or alcohol consumption, handedness). Data relating to performance in neuropsychological tests will be collected using the Inquisit 7.0 by Millisecond platform (https://www.millisecond.com/), a software widely used for the administration of computerized neuropsychological tests in clinical and research settings. Inquisit allows tasks to be performed with high temporal precision (milliseconds), supporting a wide range of cognitive paradigms for Windows and macOS devices, including touchscreens and systems with keyboard or mouse input. Cognitive tasks will be performed individually and in person on an HP Envy x360 PC running Windows 11. The scripts used for administration will be downloaded in English from the Millisecond Test Library (https://www.millisecond.com/download/library) and will be translated and adapted into Italian, maintaining the original experimental structure.

Assessment tools Selected tests were chosen to investigate selective alterations in cognitive functions related to brain areas whose activation was found to be altered in PAH patients in the aforementioned studies, such as the selective and sustained attention, working memory, processing speed and cognitive flexibility, inhibitory control, interference contrast, categorical abstraction, as well as learning and long-term verbal memory.

The performance of patients with PAH will be compared to that of the control group in working-memory abilities, attention (sustained, selective and information processing speed), executive-frontal functioning (categorisation, interference contrast, inhibitory control), cognitive flexibility (self-learning, behavioural regulation based on feedback), decision-making (decision regulation under conditions of uncertainty, sensitivity to reward) and verbal memory (long-term learning and recall of verbal material).

The following test were chosen:

* Iowa Gambling Task (IGT): developed by Bechara and colleagues (1994), this is a neuropsychological tool designed to assess short- and long-term decision-making in conditions of variable rewards and punishments. During administration, the subject is presented with an interface showing four virtual decks of cards (numbered 1 to 4), from which they must select a total of 100 cards using the mouse. Each card selected determines a win or loss of virtual money. Participants receive an initial virtual budget (£2000) with the aim of maximize their final gain by strategically choosing from decks that differ in terms of convenience. After each selection, the participant receives immediate visual feedback regarding the losses or gains associated with their choice, as well as their updated balance. The reward scheme provides that decks 1 and 2 ("disadvantageous") offer high immediate winnings accompanied, however, by occasional larger losses, resulting in a disadvantage in the long term; conversely, decks 3 and 4 ("advantageous") result in smaller but regular winnings, with occasional smaller losses, resulting in an advantage in the long term. A further distinction concerns the frequency of losses, which is high in decks 1 and 3 and low in decks 2 and 4. Score correction will be carried out according to the normative data of Maddaluno et al. (2022).
* Emotional Stroop Task (EST): a variant of the classic Stroop Test, developed by Smith and Waterman (2003) to assess the interference exerted by emotionally relevant material on cognitive processing speed and selective attention. This tool is frequently used to identify the presence of attentional biases related to specific emotional content. In this study, the original version will be adapted using emotionally salient words associated with PAH and the clinical experience of patients. The lists of neutral, positive, negative and colour-related words will be translated from the English version of the test. The test consists of a practice phase and a subsequent test phase. During the first phase, participants view 10 words belonging to the "Color Words" category on the screen, presented in a color that is incongruent with their semantic meaning in order to avoid congruence effects, with the possibility of immediate feedback on errors. In the test phase, five lists of words are presented, each consisting of 25 items belonging to the categories: "Words related to illness", "Neutral words", "Positive words", "Negative words" and "Color words". The words appear in the centre of the screen on a white background for a maximum of 2000 ms, interspersed with a 1000 ms pause. The task consists of focusing attention on the colour of the word beyond its semantic meaning, pressing the corresponding key on the keyboard (D = red; F = green; J = blue; K = yellow) as quickly as possible, on which colored squares have been superimposed for greater perceptual immediacy.
* The Rey Auditory Verbal Learning Test (RAVLT): validated in Italian by Carlesimo and colleagues (1995), it assesses learning and long-term verbal memory skills. The test consists of the verbal presentation of a list of 15 words, with no semantic connection between them and with different frequencies of use. In this study, the stimuli used will be the same as those in the Italian-validated version and will be presented to participants via a synthetised voice (Google Translate) at a constant speed of approximately one word per second. At the end of each presentation, the subject will be asked to repeat all the words they can remember, regardless of order. The same list is presented five times in a row, noting each time the total number of words correctly recalled and the presence of any intrusions. After 15 minutes in which the subject is engaged in visuospatial activities (specifically, the Visual Simon Task and the Wisconsin Card Sorting Test), a delayed recall test is performed, in which the subject is asked, without warning, to recall the words learned, without further exposure to the list. Scores will be corrected for age, gender and education and converted into equivalent scores based on the norms of Carlesimo et al. (1995).
* The Visual Simon Task (VST): a variant of the Simon Task specifically adapted for administration via keyboard, aimed at assessing working memory, inhibitory control and interference management skills (2004). Specifically, during the test, participants are presented with visual stimuli consisting of a colored square (red or blue), randomly positioned to the right or left of a central fixation cross. In congruent trials, subjects are required to press the button corresponding to the position of the square displayed ("A" for blue squares; "L" for red squares); in incongruent trials, however, participants must press the button opposite to the position of the stimulus. The test consists of a practice phase, structured in a maximum of three blocks of 8 trials each accompanied by feedback, during which participants must achieve at least 75% accuracy to access the next phase, otherwise the task is interrupted. The test phase consists of 20 trials evenly distributed according to the color and position of the stimuli, presented in random order and in such a way as to avoid the consecutive presentation of more than three stimuli from the same category.
* The Wisconsin Card Sorting Test (WCST): revisited by Heaton and colleagues (1993), is a neuropsychological test designed to assess categorical abstraction, working memory and cognitive flexibility. The test consists of a categorization task that requires the participant to associate, based on implicit criteria, a series of cards with one of the four cards shown at the bottom of the screen. The cards vary in color (red, green, yellow, blue), shape (triangle, star, cross, circle) and number (1 to 4 symbols). After each association, visual feedback ("correct" or "incorrect") is provided, allowing the subject to deduce the classification criterion. After 10 consecutive correct answers, the criterion is changed without warning, forcing the subject to update their strategy. The test ends after successfully completing six categories or using up the 128 available cards. The correction of scores in the variables detected (see below) will be carried out according to the reference standards proposed by Laiacona and colleagues (2000).

Setting All activities included in the protocol will be carried out in person in a dedicated space, in a quiet environment free from distractions.

Interaction between researchers and participants will include an initial briefing with an explanation of the instructions and ongoing support during the tasks, in order to ensure understanding, procedural correctness and comfort. The total duration of the session will be approximately 50 minutes.

At the end of the assessment, there will be a final debriefing session during which the participant will be given a clear and accessible explanation of the purpose of the tasks performed, the rationale behind the study and how the data collected will be used, with the opportunity to ask questions or give feedback on the experience.

Finally, participants will receive a feedback interview, during which the results of the neuropsychological assessment will be discussed and, if necessary, recommendations for further investigation will be provided.

N.B. Information regarding the study population and inclusion and exclusion criteria is available in the dedicated section.

Sample Size The proposed study has an exploratory observational design aimed at investigating the presence and characteristics of cognitive deficits in patients with PAH. Given the low prevalence of PAH in the general population (it is a rare disease) and the scarcity of data available in the literature on the association between this condition and cognitive impairment, it was not possible to perform a formal calculation of the sample size based on classical statistical parameters (power, level of significance, expected effect size).

For these reasons, therefore, the sample size will be determined pragmatically, based on:

* Availability of patients with a confirmed diagnosis of PAH at the centre involved in the study (15 to 30 in one year);
* Access to relevant clinical and cognitive data obtained through standardized neuropsychological assessments;
* Preliminary evidence from the literature, which reports samples ranging from 10 to 50 patients in similar studies on rare diseases or cognitive aspects in patients with chronic diseases.

Based on these elements, it is expected that approximately 15-20 patients will be enrolled during the recruitment period. Although this number does not allow for robust statistical inferences, it is nevertheless considered adequate for:

* Describing the cognitive characteristics of patients with PAH;
* Exploring possible correlations with clinical variables;
* Providing preliminary data useful for planning future controlled studies with greater statistical power.

Statistical analysis Data analysis will be conducted using statistical methods appropriate to the observational and case-control nature of the study. Descriptive statistics will first be calculated for socio-demographic and clinical variables, including mean, standard deviation, median, interquartile range, minimum and maximum values. For categorical or ordinal variables, absolute frequencies and percentages will be reported.

Independent samples t-tests (or equivalent non-parametric tests in case of violation of the assumption of normality) will be used to compare the two groups. Effect size indices (Cohen's d) will also be calculated to quantify the relevance of the differences found. Possible associations between cognitive performance and clinical and anamnestic variables (e.g., duration of illness, age at diagnosis, oxygen therapy, reported comorbidities) will also be explored using correlation analysis (Pearson or Spearman coefficient, depending on the distribution of the data). All statistical analyses will be conducted using dedicated software, in particular IBM SPSS Statistics (latest version available) and Excel for the preliminary exploration phases.

Expected results

Based on existing literature and hypotheses, it is expected that patients with PAH will differ significantly from healthy controls in terms of:

* Cognitive performance: Patients with PAH will show significantly lower performance than healthy controls in the domains investigated.
* Relationships with clinical variables: Within the PAH group, lower cognitive performance will be associated with longer disease duration, younger age at diagnosis, use of oxygen therapy, and presence of rheumatological or cardiovascular comorbidities.

ELIGIBILITY:
Inclusion criteria - PAH patients:

* Confirmed diagnosis of Pulmonary Arterial Hypertension
* Age ≥ 18 years;
* Ability to understand instructions and give informed consent;
* Absence of neurological and psychiatric comorbidities;
* Stable clinical condition, according to the treating physician's judgement;
* Willingness to participate in the study for the entire duration of the tests.

Inclusion criteria - Healthy controls:

* Matching for age (± 3 years), gender, manual laterality and level of education:
* No current or past organic and/or psychiatric disorders.

Exclusion criteria for both groups:

* Presence of medical, neurological or psychiatric comorbidities that could interfere with cognitive performance;
* Use of drugs known to affect cognitive function; Presence of sensory and/or motor deficits that could compromise test performance; Insufficient understanding of spoken and/or written Italian; Inability to give free and/or informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited consecutively from among those with a confirmed diagnosis of PAH admitted to the U.O. Cardiologia Riabilitativa of the IRCCS Maugeri - Milano. Healthy controls will be identified on a voluntary basis among IRCCS Maugeri staff, healthy family members of patients, or through other authorised internal channels. Participation in the study will be voluntary and subject to the signing of an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the performance of patients with PAH versus the control group in IGT scores | Baseline
  To compare the performance of the two groups on the Iowa Gambling Task (IGT), the following variables of interest will be collected and compared:
  * subjective ranking of the decks according to perceived convenience (ordinal ranking; e.g., 1-2-3-4);
  * number of advantageous choices (count);
  * number of disadvantageous choices (count);
  * Risk Index, calculated as the difference between the number of disadvantageous and advantageous choices (count).
Comparison of the performance of patients with PAH versus the control group in EST scores | Baseline
  To compare the performance of the two groups in EST scores, the following variables of interest will be collected and compared:
  * percentage of correct answers (%)
  * average reaction time for each category (ms)
  * interference bias, calculated as the difference between the average response times to each category and neutral words (ms).
Comparison of the performance of patients with PAH versus the control group in RAVLT scores | Baseline
  To compare the performance of the two groups in RAVLT scores the following variables of interest will be collected and compared:
  * number of words recalled in learning series (count)
  * number of words recalled in delayed recall series (count).
Comparison of the performance of patients with PAH versus the control group in VST scores | Baseline
  To compare the performance of the two groups in VST scores, the following variables of interest will be collected and compared:
  * accuracy of responses (%)
  * average reaction times by trial type (ms)
  * the 'Simon effect', calculated as the difference between the reaction times of incongruent and congruent trials (ms)
Comparison of the performance of patients with PAH versus the control group in WCST scores | Baseline
  To compare the performance of the two groups in WCST scores, the following variables of interest will be collected and compared:
  * number and percentage of perseverative responses, non-responses, and errors (count; %);
  * failures to maintain set (count);
  * Global Score, calculated as "number of cards used - (categories completed × 10)" (score).

SECONDARY OUTCOMES:
Explore the relationship between cognitive and clinical variables (disease duration, age at diagnosis, oxygen therapy, and reported comorbidities) in patients with PAH | Baseline
  Participants will undergo an initial collection of medical history data to verify their eligibility for the study. The information collected will include sociodemographic data (sex, age, marital status, number of children, employment status, level of education, years of schooling) and clinical data (past and recent medical history, current drug therapies, behavioural habits such as smoking and/or alcohol consumption, handedness). These data will be examined in relation to IGT, EST, VST, RAVLT and WCST scores .

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Maugeri - Milano, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No